CLINICAL TRIAL: NCT00809055
Title: Magnetic Resonance Imaging and Neurodevelopmental Outcomes in Preterm Infants Following Administration of High-Dose Caffeine - A Pilot Study
Brief Title: MRI and Neurodevelopment in Preterm Infants Following Administration of High-Dose Caffeine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-0849; R01HD057098-01 (NIH); HRPO 08-0849 (Other: Washington University in St. Louis)
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Apnea of Prematurity; Intraventricular Hemorrhage; Brain Injury
MeSH Terms: conditions — Apnea; Brain Injuries | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose caffeine (Experimental): Loading dose 40mg/kg IV caffeine citrate, followed 12 hours later by 20mg/kg IV caffeine citrate, followed 12 hours later by 10mg/kg IV caffeine citrate, followed 12 hours later by 10mg/kg IV caffeine citrate.
  Interventions: Drug: Caffeine citrate
- Standard dose caffeine (Active Comparator): Loading dose 20mg/kg IV caffeine citrate, followed 12 hours later with D5W placebo, followed 12 hours later with 10mg/kg IV caffeine citrate, followed 12 hours later with D5W placebo.
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — Caffeine to be administered as outlined to compare efficacy of different dosages.
  Other Names: Cafcit

SUMMARY:
Over the last 30 years the survival rates for babies born prematurely have improved greatly with research. As these babies grow up, we have found that many of the premature babies have learning and movement problems. The purpose of this research is to learn why premature infants are at risk for learning disabilities and movement problems later in childhood and whether this is changed by caffeine therapy. Caffeine is often used in premature babies to help them to breathe on their own. Nearly all babies born before 30 weeks gestation receive caffeine while they are in the neonatal intensive care unit (NICU). Scientists have shown that caffeine therapy given to premature babies reduces their disabilities.

We will use brain monitoring, including electro-encephalogram (EEG) and magnetic resonance imaging (MRI) to understand how the brain of a premature baby develops and whether caffeine in high doses enhances protection of the developing brain. Just as we monitor the heart and lungs to improve our care of premature babies, we wish to monitor the brain so that we can understand how to improve our care for the brain.

DETAILED DESCRIPTION:
Apnea is defined as a cessation of breathing for twenty seconds or greater, or as a brief episode if associated with bradycardia, cyanosis, or pallor. Recurrent apnea of prematurity occurs in up to 85% of infants born under 1000g. Standard treatment of care for apnea of prematurity is the administration of methylxanthines, specifically caffeine citrate, as a respiratory stimulant. This class of pharmacotherapy is a nonselective inhibitor of adenosine receptors. Adenosine inhibits respiratory neural output both directly and through interactions with another inhibitor of respiratory control, GABA. Adenosine A1 receptors are also thought to play a role in hypoxia-induced brain injury, and features of perinatal white matter injury have been observed in rodents treated with A1AR agonists during early postnatal life. By inhibiting adenosine effects, caffeine may play a role in preventing white matter injury. Recently, caffeine therapy for apnea of prematurity has been shown to improve the rate of survival without neurodevelopmental disability at 18 to 21 months, reduce the incidence of cerebral palsy, and reduce the incidence of cognitive delay in infants with very low birth weight.

In the last five years, multiple trials have studied the effects of using higher doses of caffeine citrate in the treatment of apnea of prematurity. Steer compared the efficacy of three dosing regimens of caffeine citrate (3, 15, and 30 mg/kg) and found that higher doses of caffeine correlated with less documented apnea and less time with oxygen saturations <85%. The effectiveness of higher caffeine doses was confirmed when Scanlon showed that a loading dose of 50 mg/kg of caffeine citrate is more effective in reducing apneic episodes within eight hours than a caffeine citrate loading dose of 25 mg/kg. Studies evaluating the long-term neurologic effects of higher doses of methylxanthines, however, have resulted in conflicting conclusions. For patients at 12 months of corrected gestational age, Steer found a higher incidence of major disabilities in the low dose caffeine group compared with the high-dose group (18% to 7.5%). Conversely, Davis reported a higher incidence of cerebral palsy in 14 year old children with birth weight below 1501g who were treated with theophylline in the newborn period than prematurely born infants without methylxanthine treatment (13% to 1.6%).

Recent advances in magnetic resonance imaging (MRI) have allowed for new techniques in visualizing brain injury and development in preterm infants by non-invasive means. Diffusion tensor imaging (DTI) is a modality of MRI that measures the translational motion of water within tissue, or "apparent diffusion." If the direction of diffusion is hindered more in one direction than another, the water motion is considered anisotropic. Water apparent diffusion in mature white matter is highly anisotropic; the directionally averaged water apparent diffusion coefficient (ADC) has been referenced at 1.0-2.0 x 10^-3 mm2/s for the infant brain, 0.8 x 10^-3 mm2/s for the adult brain. Normative values obtained by DTI have been shown to be a sensitive indicator for white and gray matter development and complexity. Both Dyet and Woodward have been able to correlate abnormal white matter signals on brain MRI in preterm infants with subsequent impairment in cognitive, motor, and neurosensory outcomes.

As caffeine use in the CAPT study has been demonstrated in low doses commenced around 3 days of life to have a positive impact on neurodevelopmental outcomes at 18 to 21 months, it would be beneficial to understand the effects of a higher dose of caffeine on both short- and long-term outcomes with an emphasis on the prevention of brain injury (intraventricular hemorrhage and white matter injury) and the improvement of neurodevelopmental development.

Thus, we propose a randomized controlled trial of high-dose versus standard low-dose caffeine therapy postulating that high doses of caffeine citrate will have beneficial effects on both short- and long-term neurologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants from 24 to 30 weeks completed PMA admitted to the neonatal intensive care unit (NICU) at St. Louis Children's Hospital. The estimated post menstrual age will be provided by the obstetrical records and compared with a Dubowitz exam at admission. The provided PMA will be used unless the Dubowitz exam has a discrepancy of greater or equal to 2 weeks, where then the Dubowitz age will be used.
* Infants must be recruited within the first 24 hours of life.

Exclusion Criteria:

* Infants over 30 weeks gestation.
* Infants who are moribund with severe sepsis, in respiratory failure, or have severe brain injury present in the first 24 hours of life. This would be defined as physiologic instability requiring >80% FiO2 for 6 hours and/or more than 2 inotropic drugs (excluding hydrocortisone), or in the attending or recruiting physicians' opinion the infant is likely to die within 24 hours or would not tolerate any handling for the protocol.
* Infants must not have received any doses of caffeine citrate prior to enrollment.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrie Inder, MBChB, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Started | 37 | 37
Completed | 28 | 30
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Caffeine | Standard Dose Caffeine | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Reported as weeks of gestational age at birth
  weeks | 26.3 (1.9) | 26.8 (1.8) | 26.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 19 | 24 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 23 | 41
  White | 17 | 12 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: White Matter Microstructural Maturation
Description: Apparent diffusion coefficient is a measure of microstructural maturation obtained from brain MRI.
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Population: 12 patients excluded from high-dose group (7 died, 2 withdrew, 3 insufficient image quality). 10 patients excluded from standard-dose group (5 died, 1 transferred, 1 parent refused MRI, 3 insufficient image quality).
Measure: Mean (Standard Deviation); unit: apparent diffusion coefficient
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 25 | 27
apparent diffusion coefficient | 1.43 (0.07) | 1.42 (0.09)

2. Secondary Outcome: Mortality Rates
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 37 | 37
participants | 7 | 5

3. Secondary Outcome: Cerebellar Hemorrhage
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 28 | 30
participants | 10 | 3

4. Secondary Outcome: Length of Time Requiring Invasive Respiratory Support
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 37 | 37
days | 4 [1 to 22] | 3 [1 to 22]

5. Secondary Outcome: Rates of Chronic Lung Disease
Description: Defined as oxygen requirement at 36 weeks PMA
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 37 | 37
participants | 19 | 18

6. Secondary Outcome: Rates of Necrotizing Enterocolitis
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 37 | 37
participants | 6 | 5

7. Secondary Outcome: Rates of Retinopathy of Prematurity
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 37 | 37
participants | 2 | 4

8. Secondary Outcome: Evaluation of EEG Seizure Burden
Description: For the first 72 hours of life, infants were monitored for seizures using continuous limited channel aEEG. Seizures were defined as a series of sharp waves, at least ten seconds in duration, which evolve in frequency, amplitude, and morphology over time and are clearly distinguishable from the background or artifact.
Time Frame: First 72 hours of life
Population: 7 patients excluded from high-dose group and 8 from standard-dose group due to recordings < 6 hours or corrupt data files.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 30 | 29
seconds | 48.9 (97.1) | 170.9 (413.1)

9. Secondary Outcome: Infant Neurobehavioral Scoring by Dubowitz Scale Prior to Discharge
Description: The Dubowitz Neurologic Examination is a standardized neurologic examination for infants at term age. It includes 6 compound optimality scores summed to obtain the total optimality score. Compound optimality scores include tone (range 0-10), tone pattern (range 0-5), reflexes (range 0-6), movements (range 0-3), abnormal signs (range 0-3), and behavior (range 0-7). The range for the compound optimality score is 0 - 34, with scores between 30.5 and 34 considered optimal and scores below 30.5 considered suboptimal.
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks
Population: 9 patients excluded from high-dose group (7 died, 2 withdrew). 6 patients excluded from standard-dose group (5 died, 1 transferred).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 28 | 31
scores on a scale | 17.4 (5.1) | 18.7 (4.3)

10. Secondary Outcome: Bayley Scales of Infant Development Cognitive Score at 2 Years of Age
Description: The cognitive portion of the Bayley Scales of Infant Development assesses development in infants and toddlers between the ages of 0 and 3 years. Raw scores are converted to scale scores. A scale score of 100 is designed to represent the population mean. Scores below 100 represent developmental delay relative to the mean and scores above 100 represent advanced development relative to the mean.
Time Frame: 2 years
Population: 13 patients excluded from high-dose group (7 died, 2 withdrew, 2 we were unable to contact, 2 did not comply with scheduled appointments). 15 patients excluded from standard-dose group (5 died, 2 withdrew, 5 we were unable to contact, 3 did not comply with scheduled appointments).
Measure: Mean (Standard Deviation); unit: score
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Number analyzed (Participants) | 24 | 22
score | 85.6 (11.6) | 88.0 (8.4)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, an average of 12 weeks.
Description: Although we detected a higher incidence of cerebellar hemorrhage in the high dose caffeine group, we have not included this outcome measure as an adverse event as it was not identified a priori. This outcome is included in the results section.
Arm/Group | High Dose Caffeine | Standard Dose Caffeine
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No